CLINICAL TRIAL: NCT05091047
Title: A Pilot Evaluation of the Effect of the Erchonia® EVRL OTC™ for the Relief of Diabetic Peripheral Neuropathy Foot Pain
Brief Title: Effect of the Erchonia® EVRL OTC™ for the Relief of Diabetic Peripheral Neuropathy Foot Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erchonia Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R-DPN-OTC Pilot
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Results first posted 2022-06-06 (Actual); Last update posted 2022-06-06 (Actual); Status verified 2022-05

CONDITIONS: Neuropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Erchonia EVRL (Experimental): 635 nanometers (nm) and 405 nm laser application
  Interventions: Device: Erchonia EVRL

INTERVENTIONS:
Device: Erchonia EVRL — 42 procedure administrations with the Erchonia® EVRL™ administered by the subject at home: Twice daily procedure administrations for 3 weeks.

SUMMARY:
This study is to see if applying red and violet low-level laser light can help to reduce foot pain associated with diabetic peripheral neuropathy,

DETAILED DESCRIPTION:
The purpose of this study is to determine whether low level laser therapy is effective in the reduction of foot pain associated with diabetic peripheral neuropathy, when used at home by non-medical professionals.

ELIGIBILITY:
Inclusion Criteria:

* Previously diagnosed with diabetes-induced Peripheral Neuropathy by a qualified health Physician.
* Over the age of 18 years of age
* Able to read and write English.
* Constant feet pain on-going over at least the past 3 months.
* Subject is willing and able to refrain from consuming any OTC and/or prescription medications including muscle relaxants and/or herbal supplements and/or recreational and medical drugs including cannabis intended for the relief of pain and/or inflammation throughout the course of study participation, except for the study-specific pain relief medication of OTC Tylenol.
* Subject is willing and able to refrain from engaging in any non-study procedure therapies for the management of foot pain throughout the course of study participation, including conventional therapies such as physical therapy, occupational therapy and hot or cold packs, as well as alternative therapies such as chiropractic care and acupuncture.
* Self-reported foot pain on the Numerical Rating Scale (NRS) is 50 or greater

Exclusion Criteria:

* Pregnant or think you might be pregnant.
* Open wounds (sores, cuts, ulcers, etc) around the feet
* Cancerous growths around the feet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Erchonia, Melbourne, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Erchonia EVRL
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Erchonia EVRL
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 3
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Duration of Feet Pain [Number; unit: years] | 6.5

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Numerical Rating Scale (NRS)
Description: The Numerical Rating Scale (NRS) assesses the level or degree of pain. With '0: no pain at all' and '100: worst pain imaginable. The subject will be asked to rate the level of foot pain he or she is experiencing at that time.
Time Frame: Baseline and 3 week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Erchonia EVRL
Number analyzed (Participants) | 8
units on a scale | 43.75 (20.98)

ADVERSE EVENTS:
Time Frame: 7 Weeks
Arm/Group | Erchonia EVRL
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/47/NCT05091047/Prot_001.pdf